CLINICAL TRIAL: NCT05580211
Title: The Clinical and Functional Imaging Effects of Non-invasive Neuromodulation on Illness Awareness in Schizophrenia
Brief Title: Neuromodulation for Schizophrenia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Scion NeuroStim (Industry)
Collaborators: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SNS-SCZ-001
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Schizophrenia
Keywords: neuromodulation
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: During the Phase I, all participants are randomized to one of two treatment stimulation patterns. In Phase II, all participants will receive the same treatment pattern.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (3):
- Investigational Stimulation Pattern 1-Randomized (Other)
  Interventions: Device: Non-invasive brainstem modulation device (stimulation Randomized)
- Investigational Stimulation Pattern 2-Randomized (Other)
  Interventions: Device: Non-invasive brainstem modulation device (stimulation Randomized)
- Investigational Stimulation Pattern-Open Label (Other)
  Interventions: Device: Non-invasive brainstem modulation device (stimulation-Open Label)

INTERVENTIONS:
Device: Non-invasive brainstem modulation device (stimulation Randomized) — Study participants will receive ~19-minute treatments twice daily in the clinic setting over 4 weeks using a non-invasive brainstem modulation device.
  Arms: Investigational Stimulation Pattern 1-Randomized; Investigational Stimulation Pattern 2-Randomized
Device: Non-invasive brainstem modulation device (stimulation-Open Label) — Study participants will receive ~19-minute treatments twice daily in the clinic setting over 8 weeks using a non-invasive brainstem modulation device.
  Arms: Investigational Stimulation Pattern-Open Label

SUMMARY:
Our proposed study employs a novel approach to determine the clinical and functional imaging effects of brainstem neuromodulation, with an investigational study device, on illness awareness in schizophrenia - a significant contributor to medication non-adherence and poor treatment outcomes, and arguably the most treatment resistant manifestation of the disorder.

The study device under investigation provides a safe and non-invasive method of brainstem stimulation that will be used in conjunction with a neuroimaging biomarker to measure brain changes associated with treatment and illness awareness.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female inpatients or outpatients ≥ 18 years of age
2. Having a DSM-V diagnosis of schizophrenia or schizoaffective disorder
3. Voluntary and capable of consenting to participation in the research study
4. Fluent in English
5. Moderate-to-severe lack of illness awareness ≤7 on the VAGUS-SR, which corresponds to a rating of ≥3 on PANSS G12 Insight and Judgment item
6. On a stable dose of antipsychotic and other concomitant medications for at least 2 months, and unlikely to undergo changes in dose during the study

Exclusion Criteria:

1. Unwilling or unable to consent to the study
2. Use of hearing aids or cochlear implants, chronic tinnitus, temporomandibular joint disease
3. Had eye surgery within the previous three (3) months
4. Ear surgery within 6 months prior to entering the study
5. Active ear infection or perforated tympanic membrane
6. Diagnosis of vestibular dysfunction
7. Unstable medical illness or any concomitant major medical or neurological illness, including a history of cardiovascular disease and seizures
8. Acute suicidal and/or homicidal ideation
9. Formal thought disorder rating ≥4 on PANSS item P2
10. DSM-V substance dependence (except caffeine and nicotine) within one month prior to entering the study
11. Positive urine drug screen at the screening visit
12. Metal implants or a pacemaker that would preclude the MRI scan
13. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Illness Awareness | 4 weeks from baseline to end of treatment
  functional MRI paradigm. The paradigm consists of a bank of brief questions or statements to which participants respond either "yes/agree" or "no/disagree". The brief statements are derived from four categories: general illness awareness, symptom awareness and attribution, awareness of need for treatment, and illness independent/control.

SECONDARY OUTCOMES:
Examine changes in brain network activity | 4 weeks from baseline to end of treatment
  functional MRI blood oxygen level dependent (BOLD) in response to an illness awareness task pre- and post-treatment. This will serve as a biomarker to rigorously test whether repeated treatment engages the posterior parietal area of the brain associated with illness awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada